CLINICAL TRIAL: NCT05945966
Title: Effects of Bilateral Versus Unilateral Lower Limb Training on Balance and Gait Parameters in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0210
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Stroke, Ischemic; Balance; Distorted; Gait, Hemiplegic
Keywords: Stroke, Ischemic; Balance; Distorted; Gait, Hemiplegic
MeSH Terms: conditions — Ischemic Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: patients will be allocated to intervention groups by randomization Patients in group A will be given MRP and PNF techniques to involve side Patients In group B will be given exercises same as above but on unaffected side.The strengthening exercises also given to this group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In this group stroke patients will be undergone task-oriented approach using motor relearning program (MRP) and proprioceptive neuromuscular facilitation (PNF) for the hemi-paretic side
  Interventions: Other: Unilateral training group (UTG)
- control group (Active Comparator): In this group stroke patients will be undergone strength training using frequency, intensity, type, time (FITT) principle to non-hemi-paretic side and task-oriented approach using motor relearning program (MRP) and proprioceptive neuromuscular facilitation (PNF) to hemi-paretic side
  Interventions: Other: Bilateral training group (BTG).

INTERVENTIONS:
Other: Unilateral training group (UTG) — stroke patients will be undergone task-oriented approach using motor relearning program (MRP) and proprioceptive neuromuscular facilitation (PNF) for the hemi-paretic side
  Arms: experimental group
Other: Bilateral training group (BTG). — stroke patients will be undergone strength training using frequency, intensity, type, time (FITT) principle to non-hemi-paretic side and task-oriented approach using motor relearning program (MRP) and proprioceptive neuromuscular facilitation (PNF) to hemi-paretic side
  Arms: control group

SUMMARY:
To determine the effects of bilateral versus unilateral lower limb training on balance and gait parameters in stroke patients

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of bilateral versus unilateral lower limb training on balance and gait parameters in stroke patients. The randomized controlled trial will recruit the stroke patients will be selected and randomly divided into two groups: Group A (unilateral training group (UTG)) and Group B (bilateral training group (BTG)).

Patients in Group A will undergo approach-oriented training using the motor relearning program (MRP) and proprioceptive neuromuscular facilitation (PNF) for the affected side, while those in Group B underwent strength training for the lower-limb muscles using Delorme's principle for the unaffected side and approach-oriented training using the MRP and PNF for the affected side for a period of six weeks, five days per week. A strengthening regimen will designed for the unaffected side, considering the frequency, intensity, time, and type (FITTs) principle provided by the American College of Sports Medicine (ACSM). The static and dynamic balance along with gait parameters will measure using the functional reach test (FRT), one-leg stance test (OLST), Berg balance scale (BBS) Dynamic Gait Index (DGI), gait parameters (stride length, gait velocity, and cadence), and Brunnstrom recovery stages (BRS) at the baseline and post rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable patients (the diagnosis was made by neurologist).
* Cognitive level is greater than 25 on MMSE.
* Chronic stroke Patients (ischemic and hemorrhagic) (6 months to 2 years).

Exclusion Criteria:

* Transient ischemic attack.
* Patients with other neurological condition, orthopedic problems, and uncontrolled metabolic disease.
* Severe hearing and visual loss.
* Uncontrolled arterial hypertension.
* Recurrent Stroke.
* Patient diagnosed with brainstem stroke and middle cerebral artery stroke.
* Patient with any cardiovascular unstable condition.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Functional reach test (FRT): | 9 months
  Functional reach test (FRT):
  It is clinical outcome measure tool for ascertaining dynamic balance in one task. It is performed with the participants in standing. It is the measure of the difference, in centimeters, between arm's length with arm at 90 degree flexion and maximum forward reach using a fixed base of support. It has 100% reliability and 76% sensitivity
Dynamic gait index (DGI): | 9 months
  Dynamic gait index (DGI):
  The DGI tests the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions. It is a useful test in individuals with vestibular and balance problems and those at risk of falls. It has high validity and reliability.
Berg balance scale (BBS): | 9 months
  Berg balance scale (BBS):
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. Its reliability is 0.98

CONTACTS AND LOCATIONS:
Overall Officials: Zeest Hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CY, Miyoshi S, Chen CH, Lee KC, Chang LC, Chung JH, Shi HY. Walking ability and functional status after post-acute care for stroke rehabilitation in different age groups: a prospective study based on propensity score matching. Aging (Albany NY). 2020 Jun 1;12(11):10704-10714. doi: 10.18632/aging.103288. Epub 2020 Jun 1. PMID 32482912
- [Background] Stoykov ME, Heidle C, Kang S, Lodesky L, Maccary LE, Madhavan S. Sensory-Based Priming for Upper Extremity Hemiparesis After Stroke: A Scoping Review. OTJR (Thorofare N J). 2022 Jan;42(1):65-78. doi: 10.1177/15394492211032606. Epub 2021 Jul 26. PMID 34311607
- [Background] Park C, Son H, Yeo B. The effects of lower extremity cross-training on gait and balance in stroke patients: a double-blinded randomized controlled trial. Eur J Phys Rehabil Med. 2021 Feb;57(1):4-12. doi: 10.23736/S1973-9087.20.06183-3. Epub 2020 Sep 6. PMID 32891079